CLINICAL TRIAL: NCT04718168
Title: GORE® ENFORM Biomaterial Product Study: A Study to Describe Multi-use Biomaterial Performance in Hernia Patients
Brief Title: GORE® ENFORM Biomaterial Product Study
Acronym: ENF 18-06
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENF 18-06
Record Dates: First submitted 2020-08-24; First posted 2021-01-22 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hernia, Ventral; Hernia, Hiatal; Hernia, Diaphragmatic; Incisional Hernia
Keywords: hernia; ventral; hiatal; diaphragmatic; incisional; mesh; Gore; W.L. Gore; Enform
MeSH Terms: conditions — Hernia, Ventral; Hernia, Hiatal; Hernia, Diaphragmatic; Incisional Hernia; Hernia; Surgical Wound | interventions — Infusions, Parenteral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Ventral/Incisional Hernia - Preperitoneal ENFORM Biomaterial (Experimental)
  Interventions: Device: Gore ENFORM Biomaterial (Preperitoneal)
- Ventral/Incisional Hernia - Intraperitoneal ENFORM Biomaterial (Experimental)
  Interventions: Device: Gore ENFORM Biomaterial (Intraperitoneal)
- Hiatal/Diaphragmatic Hernia - Preperitoneal ENFORM Biomaterial (Experimental)
  Interventions: Device: Gore ENFORM Biomaterial (Preperitoneal)
- Hiatal/Diaphragmatic Hernia-Intraperitoneal ENFORM Biomaterial (Experimental)
  Interventions: Device: Gore ENFORM Biomaterial (Intraperitoneal)

INTERVENTIONS:
Device: Gore ENFORM Biomaterial (Preperitoneal) — ENFORM Biomaterial bioabsorbable hernia mesh
  Arms: Hiatal/Diaphragmatic Hernia - Preperitoneal ENFORM Biomaterial; Ventral/Incisional Hernia - Preperitoneal ENFORM Biomaterial
Device: Gore ENFORM Biomaterial (Intraperitoneal) — ENFORM Biomaterial bioabsorbable hernia mesh
  Arms: Hiatal/Diaphragmatic Hernia-Intraperitoneal ENFORM Biomaterial; Ventral/Incisional Hernia - Intraperitoneal ENFORM Biomaterial

SUMMARY:
A prospective, retrospective, non-randomized, multicenter study with two independent hernia study cohorts (Ventral / Incisional Hernia Repair and Diaphragmatic / Hiatal Hernia Repair). The primary objective of this study is to collect GORE® ENFORM Biomaterial product commercial-use data on device functional performance and short-term patient experience.

DETAILED DESCRIPTION:
A prospective, retrospective, non-randomized, multicenter study with two independent hernia study cohorts (Ventral / Incisional Hernia Repair and Diaphragmatic / Hiatal Hernia Repair). The primary objective of this study is to collect GORE® ENFORM Biomaterial product commercial-use data on device functional performance and long-term follow up.

ELIGIBILITY:
Pre-procedure Inclusion Criteria:

The subject is / has:

1. At least 18 years old at the time of informed consent. Minimum age required by state regulations (as applicable).
2. An expected scored Class I (Clean) surgical wound using CDC Surgical Wound Classification system.
3. A planned implant with GORE® ENFORM Biomaterial for a single site ventral or hiatal hernia repair as suture line reinforcement.
4. An expected scored Grade 1 or Grade 2 using the Ventral Hernia Working Group Grading system.
5. Willing to provide informed consent and comply with follow-up requirements.

Pre-procedure Exclusion Criteria:

The subject is / has:

1. Treated in another drug or medical device study within 1 year of study enrollment.
2. Implanted with GORE® ENFORM Biomaterial in the reconstruction of cardiovascular defects.
3. Hernia repair expected to be performed as part of a bridged procedure (i.e., expected inability to perform primary closure of fascia or crura, patients requiring permanent support from the device).
4. A BMI >40.
5. Evidence of a systemic infection.
6. Cirrhosis or undergoing dialysis.
7. A wound-healing disorder.
8. Immunocompromised such as, with HIV or transplant, or receiving chemo or radiation therapy.
9. Expected to undergo mesh implantation in conjunction with any bariatric procedure and / or panniculectomy procedure.
10. A stoma.
11. Co-morbid conditions that may limit their ability to comply with study and follow-up requirements.
12. Positive pregnancy or lactation status as confirmed by site standard of care.
13. Hernias requiring treatment within multiple body regions or expected use of multiple hernia mesh devices.

Post-procedure Inclusion Criteria

At the time of index procedure, the subject is / has:

1. At least 18 years old. Minimum age required by state regulations (as applicable).
2. Implanted with GORE® ENFORM Biomaterial for a single site ventral or hiatal hernia repair as suture-line reinforcement on or before 365 days prior to site protocol amendment 3 approval date.
3. Unless there is an Informed Consent waiver issued by the Institutional Review Board (IRB), an Informed Consent Form (ICF) signed by subject.

Post-procedure Exclusion Criteria

At the time of index procedure, the subject is / has:

1. Treated in another drug or medical device study within 1 year of study enrollment.
2. Implanted with GORE® ENFORM Biomaterial in the reconstruction of cardiovascular defects.
3. Hernia repair that was performed as part of a bridged procedure (i.e., inability to perform primary closure of fascia or crura, patients requiring permanent support from the device).
4. A BMI >40.
5. Evidence of a systemic infection.
6. Cirrhosis or undergoing dialysis.
7. A wound-healing disorder.
8. Immunocompromised such as, with HIV or transplant, or receiving chemo or radiation therapy.
9. Underwent mesh implantation in conjunction with any bariatric procedure and / or panniculectomy procedure.
10. A stoma.
11. Co-morbid conditions that may limit their ability to comply with study and follow-up requirements.
12. Positive pregnancy or lactation status as confirmed by site standard of care.
13. Hernias requiring treatment within multiple body regions or expected use of multiple hernia mesh devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hernia Recurrence - Primary Device Endpoint | Through 24 months
  Clinical diagnosed hernia recurrence in the area of the initial hernia repair (within device overlap at time of index procedure).
Incidence of SSI - Primary Procedural Endpoint 1 | First Post-Procedural Visit (Days 1-45)
  Incidence of SSI, reported as a composite and individually.
Incidence of SSO - Primary Procedural Endpoint 2 | First Post-Procedural Visit (Days 1-45)
  Incidence of SSO, reported as a composite and individually.
Incidence of SSOPI - Primary Procedural Endpoint 3 | First Post-Procedural Visit (Days 1-45)
  Incidence of SSOPI, reported as a composite and individually.

SECONDARY OUTCOMES:
Freedom from potential device-related SAEs - Secondary endpoint 1 | Through 24 months
  Freedom from potential device-related Serious Adverse Events will be reported descriptively with no formal goals or hypothesis.
Re-intervention at study-treated location - Secondary Endpoint 2 | Through 24 months
  Surgical re-intervention in the area of the hernia repaired initially (e.g. drain insertion, infection, surface issues, second operation, etc.) will be reported descriptively with no formal goals or hypothesis.
Change in Quality of Life in Carolinas Comfort Scale - Secondary Endpoint 3 | Through 24 months
  For ventral hernia subjects; change in Quality of Life in Carolinas Comfort Scale as measured by a change in total score of the Carolinas Comfort Scale Quality of Life questionnaire given at follow-up visits.
  Minimum Total Score is 0 and maximum Total Score is 115. Lower score means better outcome.
Relief from GERD Symptoms - Secondary Endpoint 4 | Through 24 months
  For diaphragmatic hernia subjects; relief from GERD symptoms as measured by a decrease in the total score of the Gastroesophageal Reflux Disease Health Related Quality of Life (GERD-HRQL) questionnaire given at follow-up visits.
  Total Score: Calculated by summing the individual scores to questions 1-15. Greatest possible score (worst symptoms) = 75 Lowest possible score (no symptoms) = 0
  Heartburn Score: Calculated by summing the individual scores to questions 1-6. Worst heartburn symptoms = 30 No heartburn symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination.
  Regurgitation Score: Calculated by summing the individual scores to questions 10-15.
  Worst regurgitation symptoms = 30 No regurgitation symptoms = 0 Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (9):
- United States (9):
  - University of California - San Diego, San Diego, California
  - Institute of Esophageal and Reflux Surgery, Denver, Colorado
  - Sarasota Memorial HealthCare System, Sarasota, Florida
  - Northshore University Health System Research Institute, Evanston, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Atrium Health, Charlotte, North Carolina
  - Prisma Health - Upstate, Greenville, South Carolina
  - University of Texas Health Science Center at Houson, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No